CLINICAL TRIAL: NCT06560229
Title: Giving Resources to lOw-income Children to Enhance RecoverY
Acronym: GROCERY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2024-0466
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Discharged Pediatric Patients and Their Families

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Monthly $100 grocery gift cards for 12 months
  Interventions: Other: Grocery gift card
- Standard of Care (No Intervention): Can receive in-hospital social work referral if determined appropriate by clinical care team (also true for intervention group)

INTERVENTIONS:
Other: Grocery gift card — Monthly $100 grocery gift cards for 12 months
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to learn if an intervention to provide food support to families who are part of a Medicaid Accountable Care Organization will provide benefits. The main question it aims to answer:

Does this monthly food support intervention reduce food insecurity and healthcare utilization in these patients.

Participants will complete surveys in the hospital, 14-days after discharge, and then quarterly for up to 18 months. Families randomized to the intervention group will receive monthly grocery gift cards for one year.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a pediatric patient admitted to one of two units at our hospital with HealthVine insurance

Exclusion Criteria:

* Previous study participation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Reutilization | 30-days after discharge, 90-days after discharge, and quarterly after discharge up to 20 months
  Validated measure of reutilization which includes unplanned readmission, return to the emergency department, or a visit to urgent care
UDSA 6-question food insecurity survey | 14-days after discharge, 90-days after discharge, and quarterly after discharge up to 20 months
  Adapted version of the UDSA 6-question food insecurity survey

SECONDARY OUTCOMES:
Primary Care Healthcare Utilization | 30-days after discharge, 90-days after discharge, and quarterly after discharge up to 20 months
  Planned and unplanned visits to primary care provider
Vaccine uptake at primary care clinic | 30-days after discharge, 90-days after discharge, and quarterly after discharge up to 20 months
  Immunization percentage as part of the Medicaid accountability measure
Recovery and return to normal routine | 14-days after discharge
  Family-designed measure of recovery and return to normal routine
Post-Discharge Difficulty Coping Scale | 14-days after discharge
  Post-Discharge Coping Difficulty Scale uses an 11 point scaling format (0-10) with total scores ranging from 0 to 100. Higher scores represent greater coping difficulty.
Ability to pay for medications | 14-days after discharge, 90-days after discharge, and quarterly after discharge up to 20 months
  Family-designed measure of difficulty obtaining medications after discharge
Perceived Stress Scale | 14-days after discharge, 90-days after discharge, and quarterly after discharge up to 20 months
  Perceived Stress Scale (PSS) uses a 5 point scaling format (0-4) with total scores ranging from 0 to 40. Higher scores represent higher perceived stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No